CLINICAL TRIAL: NCT07185412
Title: Spanish Registry of Redo Procedures Following Pulmonary Vein Ablation by Pulsed Field Ablation Technology: RESET-PFA
Acronym: RESET-PFA
Status: Not yet recruiting | Type: Observational
Sponsor: Instituto de Investigación Sanitaria Aragón (Other)
Responsible Party: Principal Investigator, Javier Ramos Maqueda, Chief of the Arrhythmia Unit at Lozano Blesa University Clinical Hospital, Instituto de Investigación Sanitaria Aragón
Other Study IDs: PI24/545
Record Dates: First submitted 2025-07-09; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Cardiac Arrhythmia; Atrial Fibrillation; Pulsed Field Ablation
Keywords: Pulsed Field Ablation; Atrial fibrillation; Pulmonary vein isolation; Redo procedure; Mapping system
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- AF ablation: Patients with standard indications to AF ablation
  Interventions: Device: Pulsed Field ablation: Ablation to treat atrial fibrillation

INTERVENTIONS:
Device: Pulsed Field ablation: Ablation to treat atrial fibrillation — Pulsed Field Ablation

SUMMARY:
RESET-PFA is a prospective, multicenter, non-randomized post-market study. All patients will be treated according to the standard care followed by each center. The protocol requires enrollment of consecutive patients from each center, according to eligibility criteria. During the 12 months follow-up period, clinical atrial fibrillation recurrence, occurrence of all kinds of atrial arrhythmias and of all Adverse Events in the study population will be collected.

The purpose of this study is to prospectively evaluate during time a large population of patients with an indication for ablation of AF, collecting data on procedural success in the acute and medium- to long-term follow-up. The primary objective of the study is the determination of up to 10 clinical and procedural parameters predicting a repeat ablation procedure after the blanking period in patients that had undergone an AF ablation with pulsed field ablation through a standard of care pathway.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common sustained cardiac arrhythmia in clinical practice in the Western world, significantly impacting patient morbidity and mortality. Catheter ablation, specifically pulmonary vein isolation, has become the treatment of choice for rhythm control in patients with drug-refractory AF. Historically, thermal therapies such as radiofrequency (RF) and cryoablation have been used for pulmonary vein isolation. However, numerous studies have shown that a portion of AF recurrences pulmonary vein ablation can be attributed to pulmonary vein reconnections, suggesting suboptimal lesion durability. Pulsed field ablation (PFA), a novel non-thermal ablation technique using high-voltage, short-duration electrical pulses, has emerged as a promising alternative. PFA induces myocardial cell death via irreversible electroporation, achieving pulmonary vein isolation. Initial clinical trials demonstrated PFA's efficacy, efficiency, and safety, with favorable rates of durable pulmonary vein isolation at 3 months post-ablation.

Following commercialization and widespread adoption, multicenter registries have further confirmed PFA's efficacy and safety. Comparative studies have suggested superior long-term pulmonary vein isolation rates with PFA compared to conventional thermal therapies. Consequently, PFA has the potential to improve lesion durability and clinical outcomes for AF patients. While several studies have investigated pulmonary vein isolation durability in redo procedures in patients with clinical recurrences after PFA, results have been variable (isolation durability range: 63% - 71%), and more data is needed to fully understand the patterns of reconnection.

To our knowledge, all previous studies primarily focused on PFA during the technology's early stages and operator learning curves, potentially biasing results towards suboptimal isolation rates due to inexperience. Additionally, most studies were retrospective and single-center, with only one multicenter registry involving seven hospitals. Furthermore, none of these studies have analyzed the workflow of the index pulmonary vein isolation procedure to explain variations in lesion durability.

Therefore, the investigators present a multicenter, national, retrospective/prospective study of experienced operators to evaluate pulmonary vein isolation durability in patients with AF recurrences after PFA, focusing on the association between index procedure workflow and lesion durability.

The previous considerations seem to suggest the need to conduct a large multicentric registry of experienced operators aimed at observing current clinical practice. The registry should allow the analysis of clinical practice in relation to the current procedural recommendations, the observation of the type of methods and ablation workflow adopted and the reasons for the choices. The long-term follow-up of the patients would allow the estimation of the incidence of arrhythmic occurrences and the evaluation of the outcome, according to the clinical characteristics, the ablative strategy of the index procedure and the validation criteria at the end of the procedure. Furthermore, the prospective observation of a large number of patients treated in clinical practice approached with different ablation approaches would allow to evaluate lesion durability and residual pulmonary vein gaps that have a decisive weight in evaluating the real effectiveness of the therapy and the consequent ablation strategy during repeated ablation. These data could be extremely useful and could guide EPs in choosing the best treatment options.

The primary objective of the study is the determination of up to 10 independent predictors of repeated ablation procedure after the blanking-period in patients undergoing pulsed-field ablation of atrial fibrillation ablation through a standard of care pathway.

Secondary objectives of the study are: 12 months clinical success rate defined as freedom from any clinical atrial arrhythmia and the use of any Type I or Type III antiarrhythmic medication for the treatment of AF, AFL, or AT after the blanking period, rate and characteristics of repeated ablation procedures, association between additional applications (at the operator's discretion) at the index procedure on the durability of pulmonary vein isolation, association between occurrence of atrial arrhythmias and peri-procedural variables and ablation workflow at the index procedure, association between occurrence of atrial arrhythmias and ablation workflow at the repeated ablation procedure, analysis of repeat ablation procedures after an index PFA ablation with focus on lesion durability and type of arrhythmia recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an indication to a pulsed-field ablation procedure of Atrial Fibrillation according to current international and local guidelines (and future revisions), existing IFU or per physician discretion
* Patients who are willing and capable of providing informed consent, participating in all testing at an approved clinical investigational center or such consent will be provided by a legal representative, if required by local law or regulation.

Exclusion Criteria:

* Patients who are currently enrolled in another investigational study or registry that would directly interfere with the current study, except when the subject is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments
* Patients who are unwilling or unable to sign an authorization to use and disclose health information or an Informed Consent.
* Patients unavailable or not willing to complete follow up visits and examination for the duration of the study at the center.
* Life expectancy ≤ 12 months per physician judgment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients, clinically indicated for AF ablation, will be enrolled after signing an informed consent form and an authorization to use and disclose health information
Sampling Method: Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Title: Predictive Value of Procedural Workflow Parameters for Repeat Ablation | Index procedure through 12-month follow-up
  Association between specific procedural variables during the index procedure (e.g., number of PFA applications per vein, lesion validation method, total procedure time, voltage and activation map characteristics) as potential predictors of repeat ablation procedures and pulmonary vein isolation durability. Pulmonary vein isolation status will be assessed by electro-anatomical mapping systems in the repeat ablation procedure. The incidence of patients with isolated/not isolated pulmonary veins will be correlated with each procedural variable of the index procedure (number of PFA applications per vein, lesion validation method, total procedure time, voltage and activation map characteristics). All variables will be assessed individually and by multivariable logistic regression to establish odds ratio values.
Predictive Value of Baseline Clinical Characteristics for Repeat Ablation | 12 months post-index ablation
  Association individual baseline characteristics (e.g., age, sex, AF type, history of cardiac comorbidities, antiarrhythmic therapy) as potential predictors of repeat ablation procedures and pulmonary vein isolation durability. Pulmonary vein isolation status will be assessed by electro-anatomical mapping systems in the repeat ablation procedure. The incidence of patients with isolated/not isolated pulmonary veins will be correlated with baseline characteristics of the patient. All variables will be assessed individually and by multivariable logistic regression to establish odds ratio values.

SECONDARY OUTCOMES:
Percentage of patients free from any clinical arrhythmia and use of Type I or Type III antiarrhythmic medication | 12 months post-index ablation
  Proportion (%) of patients with documented arrhythmias and the use of any Type I or Type III antiarrhythmic medication for the treatment of atrial fibrillation, atrial flutter, or atrial tachycardia occurring after the 8-week post-ablation blanking period. Arrhythmias include atrial fibrillation, atrial flutter, or atrial tachycardia episodes lasting >30 seconds, detected by ECG, Holter monitor, or implantable loop recorder.
Rate of Repeat Ablation Procedure After Blanking Period | 12 months post-index ablation
  Proportion (%) of patients who undergo a repeat catheter ablation procedure for atrial arrhythmia recurrence occurring after the 8-week post-ablation blanking period. Arrhythmias include atrial fibrillation, atrial flutter, or atrial tachycardia episodes lasting >30 seconds, detected by ECG, Holter monitor, or implantable loop recorder.
Durability of Pulmonary Vein Isolation at Repeat Procedure | At time of repeat ablation (if performed within 12 months)
  Proportion of pulmonary veins (%) that remain durably isolated at the time of repeat ablation procedure due to atrial arrhythmia recurrence occurring after the 8-week post-ablation blanking period. Pulmonary veins isolation will be assessed by using high-density mapping.
Technical workflow variables of the PFA Procedure Over Time | Measured during index procedure
  This outcome aims at evaluating changes in technical periprocedural variables, such as total skin-to-skin time (from first puncture to final catheter withdrawal), catheter dwell time (from transeptal time to final catheter withdrawal), ablation time (from first PFA application to final PFA application) and fluoroscopy time (during the entire procedure) across the study period. Temporal milestones will be evaluated to reflect improvements in workflow efficiency as operator experience increases.
Electroanatomical Voltage Characteristics as Predictors of Arrhythmia Recurrence | 12 months post-index ablation
  Assessment of baseline left atrial voltage characteristics, measured as the mean electrical voltage of bipolar signals in the pulmonary veins and posterior wall healthy tissue during index procedure by using electro-anatomical mapping systems, as predictors of atrial arrhythmia recurrence after the 8-week blanking period.
Activation Map Patterns as Predictors of Predictors of Arrhythmia Recurrence. | 12 months post-index ablation
  Assessment of differential left atrial activation patterns obtained during the index procedure by means of mapping with an electro-anatomical mapping system, as predictors of atrial arrhythmia recurrence after the 8-week blanking period.
Acute lesion validation during Index Procedure as Predictor of Arrhythmia Recurrence | 12 months post-index ablation
  Assessment of whether performing or no acute lesion validation of pulmonary vein isolation, by means of entrance/exit block, or differential pacing response, during the index ablation may be a predictor of arrhythmia recurrence during follow-up.
Acute lesion validation during Index Procedure as Predictor of pulmonary vein isolation | 12 months post-index ablation
  Assessment of whether performing or no acute lesion validation of pulmonary vein isolation (by means of entrance/exit block, or differential pacing response) during the index ablation may be a predictor of pulmonary vein isolation during the repeat ablation procedure due to atrial arrhythmia recurrence occurring after the 8-week post-ablation blanking
Number of PFA applications during Index Procedure as Predictor of pulmonary vein isolation | 12 months post-index ablation
  Correlation of number of applications in each pulmonary vein, and the use of additional application at operator's discretion during the index ablation procedure, with the pulmonary vein isolation status during repeated ablation procedure due to atrial arrhythmia recurrences.
Impact of Pre-procedural Imaging on Arrhythmia Recurrence | 12 months post-index ablation
  Assessment of the percentage of patients with any pre-procedural imaging of the left atria available to guide ablation with documented arrhythmias and the use of any Type I or Type III antiarrhythmic medication for the treatment of atrial fibrillation, atrial flutter, or atrial tachycardia occurring after the 8-week post-ablation blanking period. Evaluation if the availability of any pre-procedural imaging is associated with a lower recurrence of atrial arrhythmia after ablation compared with those without previous imaging.
Number of patients with antiarrhythmic therapy discontinued after ablation compared to the baseline status. | 12 months post-index ablation
  Rate of patients (%) in which the antiarrhythmic therapy was discontinued after ablation compared to the baseline pharmacological status during the 12-month period of follow-up.
Differential evolution of AF category after ablation | 12 months post-index ablation
  Rate of patients (%) with a change in the AF typus or evolution (from paroxysmal to persistent AF; or from persistent to paroxysmal AF) registered in the repeated ablation procedure, compared to the index baseline status. AF will be recorded by ECG, Holter monitor, or implantable loop recorder.

CONTACTS AND LOCATIONS:
Locations (1):
- Unidad de Arritmias. Departamento de Cardiología. Hospital Universitario Lozano Blesa., Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No